CLINICAL TRIAL: NCT01783652
Title: Adaptation of a U.S. Internet Tool to Prevent Depression and Addiction in Hong Kong Adolescents
Brief Title: Adapted and Translated, Adolescent Depression, Internet Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: catch_it_2013
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Adolescent - Emotional Problem
Keywords: Adolescent depression; internet intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Study participants in the intervention group will be given access to an anti-depression website and have four telephone follow-up within the 1-year study period.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): Study participants in the control group will not received any depression-related service other than an interactive anti-smoking website provided by the University of Hong Kong.

INTERVENTIONS:
Behavioral: Intervention group — Participants in the intervention group will have access to the anti-depression website modified and translated by the University of Hong Kong. 10 chapters on understanding depression, identifying depression symptoms and techniques tackling depression will be covered. Exercises and built-in questionnaires on measuring emotions will be provided in the website. Additional telephone follow-up counseling at the third, sixth and twelfth months will be conducted.
  Arms: Intervention group

SUMMARY:
Objectives :

The key objective of this study is to develop new interventions that addresses the diverse needs and circumstances of Hong Kong adolescents with depressive symptoms in community settings. Collaboration between medical professionals and social workers may prevent the occurrence of depression and misguided attempts to self-treat with alcohol and / or drugs in our adolescents.

Methods :

To address this intervention gap in the United States, Dr. Van Voorhees, a research collaborator of Dr. Chim and Dr. Ip, developed and conducted a phase 2 clinical trial of a primary care internet-based depression prevention intervention (CATCH-IT, Competent Adulthood Transition with Cognitive Behavioral Humanistic and Interpersonal training). It has been observed clinically that the strategy could reduce depressed mood, increased social support and reduced depressive episodes at 12 month follow-up.

The investigators now propose to study if an adaptation of the CATCH-IT website for Hong Kong Chinese adolescents may lead to significant reductions in depressed mood. In this pilot trial, the investigators propose to test the efficacy of the Adapted and Translated version of CATCH-IT (AT-CATCH) against the placebo approach in preventing the onset of depressive episodes in a group of adolescents (aged 13-17) who have depressive symptoms, but have not developed depression yet.The case group will have access to the AT-CATCH website while the control group will only be allow to use the anti-smoking website.

The investigators hypothesize that compared to youth in the control group, youth assigned to the AT-CATCH group will have a lower hazard ratio of major depressive episodes and decreased alcohol / drug use frequency over 2 years. Moreover, compared to youth in the control group, youth in the AT-CATCH program will demonstrate a steeper slope of improved symptoms through growth curve analysis and fewer depressed days over the study period.

DETAILED DESCRIPTION:
Although efficacious psychological and pharmacological treatments for adolescent depression have been demonstrated, any single approach only helps about 50-75% of those treated. Furthermore, adolescents have low rates of care seeking, and many primary care patients find group therapy to be the least acceptable treatment for depression. Limited supply of mental health specialists make face-to-face counseling difficult to implement, hence the internet is a promising modality for the delivery of preventive interventions. Therefore, prevention of depression in at-risk adolescents may be more cost-effective and less distressing than allowing for the depressive symptoms to become more severe.

Key issues - international level:

As proposed by the World Health Organization (WHO) and National Institute of Mental Health (NIMH), prevention of mental disorders has become a major health need (9), and a primary care internet-based depression prevention intervention strategy should be developed. Such care has already been provided for depression in the U.S. by Dr. Van Voorhees, suggesting the intervention must:

1. have broad reach into at-risk populations;
2. work outside of traditional mental health systems;
3. use new technologies;
4. build on previous clinical trials;
5. reduce identified disorders/enhance functional outcomes;
6. include families; and
7. be personalized

Key issues - local level Developing new interventions that incorporate the diverse needs and circumstances of Hong Kong adolescents with depressive symptoms in community settings is our key strategic objective. While it is ideal to have a series of primary care physician consultations for at-risk adolescents, this is not available and too expensive for the lower socioeconomic class. This lack is apparent in both the East and the West. The U.S. has built up a new cost-effective prevention strategy for depression in primary care system; however, such a strategy may not be able to be incorporated into the public health sector. Hence, the collaboration between physicians and social workers will be used for this study.

Inclusion criteria:

138 adolescent participants (ages 13 to 21) who experience a moderately elevated level of depressive symptoms on the CES-D scale (score 16-34) will be recruited to join the study. Participants may or may not have had a past history of depression, anxiety and/or substance abuse.

Outcome measures to compare between 2 groups:

i) depressive episodes and symptoms Assessment of adolescent depression by the Centre of Epidemiological Studies Depression Scale (CES-D) and Depression Anxiety Stress Scale (DASS) are a standard diagnostic test for assessment of adolescent's depression. The scores of both groups would be measured and compared in 3 follow-ups to study the effect and its sustainability of the website intervention.

ii) use of alcohol and drugs Assessment of drinking and drug use behavior of adolescents by CRAFFT Screening Test, which includes questions regarding alcohol and drug use situations in the past 12 months, and additional assessment for those who show a significant problem. There are 6 questions covering road safety, drug-use habits, and influences of using drugs or alcohol.

ELIGIBILITY:
Inclusion Criteria:

* age 13 to 21
* experience a moderately elevated level of depressive symptoms on the CES-D scale (score 16-34)
* may or may not have had a past history of depression, anxiety and/or substance abuse

Exclusion Criteria:

* currently diagnosed with depression, schizophrenia, or bipolar affective disorder ;
* currently taking antidepressants or psychotropic medication ;
* CES-D score equal or higher than 35, or a proved serious medical illness that causes significant disability or dysfunction ;
* exhibit significant reading impairment, mental retardation, developmental disabilities
* serious imminent suicidal risk or other conditions that may require immediate psychiatric hospitalization
* have extreme, current drug / alcohol abuse (greater than or equal to 2 on the CRAFFT)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | 12 months
  Centre for Epidemiological Studies Depression Scale (CES-D) : at baseline, 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Depression measurement | 12 months
  Depression Anxiety Stress Scale (DASS) : at baseline, 3 months, 6 months and 12 months
alcohol abuse | 12 months
  CRAFFT Screening Test : at baseline, 3 months, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Chim, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong, China